CLINICAL TRIAL: NCT03158870
Title: Influence of Surgeon-anesthesiologist Collaboration on Patient Outcomes After Pheochromocytoma Surgery
Brief Title: Surgeon-Anesthesiologist Collaboration
Acronym: CCAP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0030
Record Dates: First submitted 2017-05-17; First posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Pheochromocytoma; Collaboration
MeSH Terms: conditions — Pheochromocytoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pheochromocytoma: Patient who underwent surgical procedure for pheochromocytoma
  Interventions: Procedure: Surgery complications

INTERVENTIONS:
Procedure: Surgery complications — Assessment of the influence of surgeon-anesthesiologist collaboration on surgery complications during and up to 30 days after pheochromocytoma surgery.

SUMMARY:
Collaboration between the surgeon and the anesthesiologist is key for delivering a safe pheochromocytoma surgery. This study aims to establish the collective performance of surgeon-anesthesiologist team by quantifying the relationship between their previous collaborations and patient complications.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent surgical procedure for pheochromocytoma in 8 French university hospitals from January 2000 to December 2016

Exclusion Criteria:

* Age < 18 years old
* Patients operated for incidentaloma or with paraganglioma diagnosis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients operated for pheochromocytoma
Sampling Method: Non-Probability Sample
Enrollment: 1122 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Presence of an intraoperative hemodynamic instability | At the time of surgery (less than 4 hours)
  An intraoperative hemodynamic instability is defined as the occurrence of at least one intraoperative episode of systolic blood pressure ≥ 160 mmHg and at least one episode of mean blood pressure ≤ 60 mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Pôle Information Médicale Evaluation Recherche des Hospices Civils de Lyon - Centre Hospitalier Lyon Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No